CLINICAL TRIAL: NCT02231814
Title: Dietary Therapy Using the Crohn's Disease Exclusion Diet (CDED) With Partial Enteral Nutrition or Alone for Induction and Maintenance of Remission in in Adults With Mild to Moderate Crohn's Disease- A Pilot Study
Brief Title: The Crohn's Disease Exclusion Diet With Partial Enteral Nutrition or Alone in Adult Patients With Crohn's Disease
Acronym: CDED-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Arie Levine (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Arie Levine, Director, Pediatric Gastroenterology and Nutrition unit., Wolfson Medical Center
Organization: Wolfson Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0105-14
Record Dates: First submitted 2014-08-27; First posted 2014-09-04 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Mild to moderate Crohn's Disease; Diet; Enteral Nutrition
MeSH Terms: conditions — Crohn Disease | interventions — penclomedine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Crohn's Disease Exclusion Diet+Partial Enteral Nutrition (PEN): Crohns Disease Exclusion Diet + PEN
  Interventions: Dietary Supplement: Crohns Disease Exclusion Diet + PEN
- Group 2 (Experimental): Crohn's Disease Exclusion Diet alone with a calcium supplement
  Interventions: Other: Crohns Disease Exclusion Diet

INTERVENTIONS:
Dietary Supplement: Crohns Disease Exclusion Diet + PEN — Patients will use the CDED for a 24 week period, coupled with 1000 m"l of polymeric formula (1 Kcal/m"L) for the first 6 weeks. For weeks 7 to 24 patients will use the CDED coupled with 600 ml formula and a calcium supplement. The CDED is divided into 3 stages: 0-6 weeks induction phase, weeks 7-12 step down phase, weeks 13-24 maintenance phase.
  Other Names: CDED + Liquid dietary formula
  Arms: Group 1
Other: Crohns Disease Exclusion Diet — Crohn's Disease Exclusion Diet alone with a calcium supplement during the study (0-24). The CDED is divided into 3 stages: 0-6 weeks induction phase, weeks 7-12 step down phase, weeks 13-24 maintenance phase.
  Other Names: CDED
  Arms: Group 2

SUMMARY:
This study will evaluate a novel diet for adult crohn's disease patients (The Crohn's Disease Exclusion Diet - CDED). Half of the patients in this study will receive the CDED alone while the other half will receive the CDED and a liquid diet formula, for 24 weeks.

DETAILED DESCRIPTION:
Environmental factors, the microbiome (bacteria in our gut) and innate immunity all play a role in the pathogenesis of Crohn's disease .Exclusive enteral nutrition (EEN) was found to be effective for inducing remission in active pediatric Crohn's disease, while Partial Enteral Nutrition (PEN) with free diet was not; suggesting that the mechanism of EEN depends on exclusion of dietary components. Dietary factors may play a role in the pathogenesis of the disease, and maybe an important under-investigated therapeutic target.

"The Crohn's Disease Exclusion Diet" (CDED) is a palatable diet excluding components suspected to interfere with the bacteria in our gut or impair immune mechanisms. Our group previously evaluated 47 patients using the Crohn's disease Exclusion Diet + 50% Polymeric formula for 6 weeks, and demonstrated a 78% response rate and 70% disease remission rate using stringent criteria. This was accompanied by a highly significant reduction in markers for inflammation (C-reactive protein (CRP) and Erythrocyte Sedimentation Rate (ESR)), and normalization of CRP in 70% of those entering remission. Among these patients were 13 adults aged 19-32, the remission rate in these 13 patients was 69%, similar to the pediatric data. Importantly, 6/7 patients in this study who refused to drink formula and just used the diet achieved remission, suggesting that the exclusion and not partial enteral nutrition are responsible for the high remission rate. Our former study did not evaluate mucosal healing as an end point, since performing colonoscopies after 6- 12 weeks of therapy is neither ethical nor feasible in children.

At present, data about nutritional therapy and this new dietary approach have been generated primarily in children, and this new diet has not been evaluated for early mucosal healing. The objectives of this pilot study are to generate data in adults, evaluate the diet over a longer period of time (24 weeks) and evaluate mucosal healing. The study is a prospective open label randomized controlled pilot trial in adults, with mild to moderate Crohn's disease who will receive the Crohn's Disease Exclusion Diet (CDED) for 24 weeks.

If effective, this could enable use of a feasible, safe intervention for induction and maintenance of remission as a new therapy or as an adjunctive therapy with medical therapy.

ELIGIBILITY:
Inclusion Criteria

1. Informed consent
2. Established Crohn's disease
3. Aged 18-55
4. Duration of disease up to 5 years
5. Harvey Bradshaw Index 5 ≤( HBI) ≤15
6. Patients with uncomplicated disease involving the terminal ileum and or cecum
7. Patients who performed colonoscopy (or MR/CTEnterography with elevated calprotectin>200) demonstrating active disease in the previous 8 weeks

Exclusion Criteria

1. Patients with severe Disease (HBI > 15) or HBI<5
2. Pregnancy,
3. Patients with active extraintestinal disease, current B2 (Fixed non inflammatory stricture1 or small bowel obstruction) or B3 disease,
4. Patients who used immunomodulator <8 weeks, or had dose changed in past 8 weeks,
5. Patients with current or past use of biologics, or use of systemic steroids2,
6. Patients with deep ulcers involving the colon distal to the splenic flexure on most recent colonoscopy
7. Any proven current infection such as positive stool cultures or positive tests for parasites or C. difficile. Stool tests are mandatory only if diarrhea is present.
8. Active Perianal disease ( clarification-fistula with discharge or abscess)
9. Patients who have undergone an intestinal resection
10. Patients with systemic disease including: type 2 diabetes, kidney failure, liver failure, neurological disease, active heart disease and patients with active autoimmune condition requiring medication3
11. Patients unwilling to consume any animal source protein (eggs, chicken or fish).

Comments:

1. Patients with ileo-cecal valve narrowing maybe included
2. Patients active despite budesonide may enter the trial if they are on 3 mg, and stop budesonide within 14 days of commencement of the trial.
3. Patients with Celiac disease or Hashimoto Thyroiditis can be enrolled

   -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Clinical remission defined as Harvey Bradshaw Index (HBI)<5 | Week 6

SECONDARY OUTCOMES:
Steroid free remission between groups | Week 6, 12 and 24.
Mucosal healing | Week 24-26
Changes in mean C-Reactive Protein (CRP) | Weeks 6, 12 and 24.
Change in mean fecal calprotectin | Week 6, 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Arie Levine, MD, Principal Investigator — Wolfson Medical Center; Iris Dotan, MD, Principal Investigator — Tel Aviv Medical Center; Irit Hermesh, MD, Principal Investigator — Rambam Medical Center,Haifa
Locations (4):
- Israel (4):
  - Haemek, Afula
  - Wolfson Medical Center, Holon
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Background] Sigall-Boneh R, Pfeffer-Gik T, Segal I, Zangen T, Boaz M, Levine A. Partial enteral nutrition with a Crohn's disease exclusion diet is effective for induction of remission in children and young adults with Crohn's disease. Inflamm Bowel Dis. 2014 Aug;20(8):1353-60. doi: 10.1097/MIB.0000000000000110. PMID 24983973
- [Background] Yanai H, Levine A, Hirsch A, Boneh RS, Kopylov U, Eran HB, Cohen NA, Ron Y, Goren I, Leibovitzh H, Wardi J, Zittan E, Ziv-Baran T, Abramas L, Fliss-Isakov N, Raykhel B, Gik TP, Dotan I, Maharshak N. The Crohn's disease exclusion diet for induction and maintenance of remission in adults with mild-to-moderate Crohn's disease (CDED-AD): an open-label, pilot, randomised trial. Lancet Gastroenterol Hepatol. 2022 Jan;7(1):49-59. doi: 10.1016/S2468-1253(21)00299-5. Epub 2021 Nov 2. PMID 34739863